CLINICAL TRIAL: NCT03269734
Title: Evaluation of the Accuracy of the Vessel Navigator (Philips Healthcare) Tool for Catheterization of Aortic Arch and Supra-aortic Vessels - ARCHIBALD
Brief Title: Evaluation of the Accuracy of the Vessel Navigator Tool for Catheterization of Supra-aortic Vessels - ARCHIBALD
Acronym: ARCHIBALD
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_RBC_2016_1
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2017-12

CONDITIONS: Vascular Diseases; Cerebrovascular Diseases; Cardiovascular Diseases; Aortic Aneurysm; Arteriovenous Malformation
Keywords: Vascular Diseases; Cerebrovascular Diseases; Cardiovascular Diseases; Aortic aneurysm; Arteriovenous malformations; Catheterization
MeSH Terms: conditions — Vascular Diseases; Cerebrovascular Disorders; Cardiovascular Diseases; Aortic Aneurysm; Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study compares the accuracy of fusion imaging (Fusion Roadmap) versus real-time X-ray imaging (Roadmap) during catheterization of supra-aortic trunks of in patients with aneurysms or arteriovenous malformations.

DETAILED DESCRIPTION:
Catheterization of is performed for the diagnosis and treatment of cerebrovascular diseases. It is performed under X-ray scopy in frontal incidence with possible variations of the angulation of the arch to optimize the visualization of vessels 'origin (brachiocephalic trunk, left and right common carotid arteries, subclavian arteries).

Before the beginning of catheterization, a conventional arterial roadmap with iodine injection is usually performed. The Vessel Navigator (VN) developed by Philips allows the use of pre-acquired angio-scan or angio-MRI image by superimposing it (X-ray Fusion) on X-ray scopy to provide the arterial tracing (Fusion Roadmap).

An angio-MRI (Philips 3 Tesla MRI) imaging of the aortic arch will be first performed (as part of preoperative assessment or systematic follow-up of aneurysms or arteriovenous malformations). A first operator will perform the arteriography under the usual conditions without using the VN. A second operator will have access to the fusion imaging and will assess the accuracy of the coregistration. Snapshots will be taken by the second operator.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative assessment or systematic follow-up of aneurysms or arteriovenous malformations, arterial cervical or intracranial stenosis, head and neck vascular tumors.

Exclusion Criteria:

* Patients with contraindication to intravenous contrast.
* Patients with catheterization of the supra-aortic vessels in an emergency settings (Stroke, acute bleeding)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with preoperative assessment or systematic follow-up of aneurysms or arteriovenous malformations, arterial cervical or intracranial stenosis, head and neck vascular tumors.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Offset (in mm) between the lateral edge of the opacified artery and that visualized with the fusion imaging. | baseline
  Measurement will be performed 1 cm above each ostium. There will be 4 measurements per patient (4 vessels analyzed).

SECONDARY OUTCOMES:
Subjective opinion of the second operator on the aspect of registration to carry out the catheterization (satisfactory or not). | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël BLANC, MD, Principal Investigator — Fondation ophtalmologique de Rothschild
Locations (1):
- Fondation Opthalmologique A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided